CLINICAL TRIAL: NCT00311818
Title: 44-week, Parallel, Open, Randomized, Multinational, Multi-center Clinical Trial to Compare Efficacy and Safety of the Combination Therapy of an Oral Anti-diabetic Drug Treatment With Either HOE901 Insulin Once Daily or Lispro Insulin Analogue at Mealtime in Type 2 Diabetes Mellitus Patients Poorly Controlled With Oral Anti-diabetic Drug Treatment.
Brief Title: Insulin Glargine in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4040
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin glargine

SUMMARY:
Primary objective:

* To compare efficacy of oral antidiabetics (OAD) combination therapy with either HOE901 insulin analogue once daily or Lispro insulin analogue at mealtime in terms of change in HbA1c (baseline to endpoint).

Secondary objectives:

* To compare the OAD combination therapy with either HOE901 insulin analogue once daily or Lispro insulin analogue at mealtime in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 Diabetes mellitus for at least 1 year (no history of ketoacidosis) and treatment with oral antidiabetics (OAD) for at least 6 months prior to study entry
* Subjects poorly controlled with previous OAD treatment: any mono or combination therapy approved in combination with insulin according to local SPCs (summary of product characteristics), not including use of alpha-glucosidase inhibitors, at a stable dose for least 3 month prior to study entry
* Poor metabolic control with HbA1c (glycosylated hemoglobin) values between 7.5 % and 10.5 % and FBG > or = 120 mg/dl (6.6 mmol/l)
* Body mass index < or = 35 kg/m2
* Ability and willingness of a tight antidiabetic therapy under a stable life-style with regular meals and to perform blood glucose self monitoring and especially blood glucose profiles using a blood glucose meter at home, as evidence by daily FBG measurements and a complete 8-point blood glucose profile obtained over a 24-hour period

Exclusion Criteria:

* Treatment with any insulin in the last 4 weeks prior to study entry
* Diabetes mellitus following pancreatectomy
* GAD positive (glutamic acid decarboxylase)
* Diabetic retinopathy with surgical treatment (laser photocoagulation or vitrectomy) in the 3 months prior to study entry or which may require surgical treatment within 3 months of study entry
* Pregnant or breast-feeding
* Women of childbearing potential who did not take adequate contraceptive protection such as systemic hormones (birth control pills, implant), intrauterine device, or a barrier method (diaphragm with intravaginal spermicidal, cervical cap, male or female condom)
* History of hypersensitivity to the study medication or to drugs with similar chemical structures
* Treatment with any investigational drug in the last 3 months before study entry
* Previous enrollment in a study involving HOE901 insulin analogue
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol (e.g. non-cardio selective beta-blockers, systemic corticosteroids)
* Clinically relevant cardiovascular, gastrointestinal, hepatic, neurologic, endocrine, hematological or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* History of drug or alcohol abuse
* Impaired hepatic function, as shown by, but not limited to,alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) above 3x the upper limit of normal, if no lower values are required by the individually administered OAD
* Impaired renal function, as shown by, but not limited to, serum creatinine > 177 mmol/l (> 2 mg/dl), if no lower values are required by the individually administered OAD

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects with HbA1c: ≤ 6.5 %, 6.5 %< HbA1c ≤ 7.0 %, 7.0 %<HbA1c ≤ 8.0 % and HbA1c > 8.0 % | at endpoint

SECONDARY OUTCOMES:
Change in fasting blood glucose, (FBG) | baseline to endpoint
Frequency of subjects with: FBG ≤ 100 mg/dl (5.5 mmol/l), 100 mg/dl < FBG ≤ 126 mg/dl(7.0 mmol/l) and FBG > 126 mg/dl (7.0 mmol/l) | at endpoint
Change in nocturnal blood glucose | baseline to endpoint
Change in fasting plasma glucose | baseline to endpoint and all visits
Change in mean daytime blood glucose | baseline to endpoint
Change in mean daily blood glucose | baseline to endpoint
Change in blood glucose at the remaining time points of the 8-point-blood glucose profiles | baseline to endpoint
Frequency of subjects with hypoglycemic events (overall, severe, nocturnal, symptomatic) | from the inform consent signature to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, Study Director — Sanofi

REFERENCES:
- [Result] Bretzel RG, Nuber U, Landgraf W, Owens DR, Bradley C, Linn T. Once-daily basal insulin glargine versus thrice-daily prandial insulin lispro in people with type 2 diabetes on oral hypoglycaemic agents (APOLLO): an open randomised controlled trial. Lancet. 2008 Mar 29;371(9618):1073-84. doi: 10.1016/S0140-6736(08)60485-7. PMID 18374840